CLINICAL TRIAL: NCT07132060
Title: MRI-guided Dose Intensification Program Locally Advanced Pancreatic Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024.174
Record Dates: First submitted 2025-08-12; First posted 2025-08-20 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Pancreatic Cancer
Keywords: MRI-guided irradiation; Dose escalation; Ultrahypofractionation
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultrahypofractionation Phase (Experimental): MR-Guided Ultrahypofractionation
  Interventions: Radiation: MR-guided Irradiation

INTERVENTIONS:
Radiation: MR-guided Irradiation — MR-guided Irradiation

SUMMARY:
The goal of this clinical trial is to learn if the use of dose-escalated MRI-guided irradiation increases the rates of disease control in patients with pancreatic cancer

DETAILED DESCRIPTION:
The implementation of Magnetic Resonance Image Guided Radiotherapy (MRgRT) into a Pancreatic Cancer Intensification Program maximizes treatment objectives rates due to the better visualization and online dose-adaptation pancreatic tumor.

Rationale In the radiation setting, MRI provides superior soft tissue contrast compared to standard onboard X-ray imaging improving inter- and intra- observer delineation variation. MRgRT offers the opportunity to adapt the plan at each fraction to the anatomical changes seen (Henke et al., 2018). This creates a much better CTV to OAR ratio in a 50Gy/5Rx scenario.

Primary Objectives A. To achieve a 1-year survival of 85%. B. To decrease grade 4-5 gastrointestinal events to less than 5%.

Secondary Objectives A. Determination of blood and urine biomarkers of treatment response and toxicity .

B. Determination of radiomics biomarkers of treatment response and toxicity . C. Determination of quality of life with the EORTC QLQ-C30 Questionnaire .

ELIGIBILITY:
Inclusion Criteria:

* Selection criteria includes patients with unresectable and borderline resectable and medically inoperable pancreatic cancer that will receive neoadjuvant chemotherapy followed by chemoirradiation.
* No prior radiation therapy to the target areas;
* Karnofsky performance status > 70 with medical condition not contraindicating treatment with radical intent including neoadjuvant chemotherapy followed by chemoirradiation.
* WBC equal or greater than 3500 mm^3; platelet count equal or greater than 135000 mm^3; hemoglobin equal or greater than 10 gr/L; BUN equal or less than 20; serum creatinine equal or less than 2.0.

Exclusion Criteria:

* Inability to undergo an MRI scan

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 2-years
  A. To achieve a 1-year survival of 85%.

SECONDARY OUTCOMES:
Adverse Events | 2-years
  To decrease grade 4-5 gastrointestinal events to less than 5%.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Martínez-Monge, M.D., Principal Investigator — Clínica Universidad de Navarra; Luis Fuertes, M.D., Principal Investigator — Clínica Universidad de Navarra

IPD SHARING:
Plan to Share IPD: Yes
On request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 5-years
Access Criteria: On request